CLINICAL TRIAL: NCT05126147
Title: A Randomized Controlled Trial on the Effect of Hydroxychloroquine in Mild Graves' Orbitopathy
Brief Title: Hydroxychloroquine in Mild Graves' Orbitopathy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202101055MINB
Record Dates: First submitted 2021-10-05; First posted 2021-11-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Graves Ophthalmopathy
Keywords: Graves' ophthalmopathy; Graves' disease; Hydroxychloroquine; Orbital volumetry; GO-QoL questionnaire
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Experimental): Hydroxychloroquine 200mg twice daily for 6 months.
  Interventions: Drug: Hydroxychloroquine
- Control (No Intervention): Observation and active surveillance.

INTERVENTIONS:
Drug: Hydroxychloroquine — Compare the effects of hydroxychloroquine 200mg twice daily for 6 months with those without treatment.
  Other Names: Plaquenil
  Arms: Hydroxychloroquine

SUMMARY:
This study is aimed to investigate the effect of hydroxychloroquine in patients with mild Graves' orbitopathy (GO).

DETAILED DESCRIPTION:
Graves' orbitopathy (GO) is one of the common manifestations of Graves' disease (GD), which results in proptosis, eyelid retraction, soft tissue swelling, diplopia or even visual acuity impairment. In addition, mental health and quality of life are often affected. In current guidelines, limited treatment options are suggested for patients with mild GO.

Recently, cell study revealed that there are multiple effects of hydroxychloroquine (HCQ) on orbital fibroblasts in patients with mild GO, including suppression of cell proliferation, adipogenesis and production of hyaluronic acid, which poses a great potential in the treatment of mild GO clinically. This randomized controlled trial is aimed to investigate the effects of HCQ in patients with mild GO on the effects of ophthalmic outcomes, quality of life, orbital volumetry on orbital computed tomography, serum inflammatory and fibrosis markers.

ELIGIBILITY:
Inclusion Criteria:

* Mild GO according European Group on Graves' orbitopathy (EUGOGO) guidelines diagnosed by endocrinologist and ophthalmologist.
* No previous treatment of GO except for eyedrops
* Euthyroidism (normalized free T4 and TSH) for at least 2 months. If radioactive iodine is used for hyperthyroidism, euthyroidism needs to be achieved for at least 6 months.

Exclusion Criteria:

* Moderate-to-sever or sight-threatening GO according to EUGOGO guidelines diagnosed by endocrinologist and ophthalmologist.
* Pregnancy
* Drug or alcohol abuse
* Unable to comply with the study protocol
* Unable to obtain informed consent
* Use of hydroxychloroquine or systemic steroid within 3 months prior to enrollment
* History of side effects of hydroxychloroquine
* History of retinopathy
* Renal dysfunction (estimated glomerular filtration rate (eGFR) < 60ml/min)
* Hepatic dysfunction (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 x upper limit)
* Anemia (hemoglobin (Hb) < 10g/dl)
* Neutropenia (absolute neutrophil count < 100/uL)
* Thrombocytopenia (platelet (PLT) < 150000/uL)
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Porphyria cutaneous tarda
* Allergy to 4-aminoquinoline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of ophthalmic outcome | at 24 weeks and 48 weeks
  The ophthalmic outcome is a composite outcome which includes three components: eyelid aperture, soft tissue involvement and exophthalmos.
  The outcome is defined as "improvement" if any of the three components improves without deterioration of any other components. The outcome of "deterioration" is defined if upgrading of soft tissue involvement or evidence of worsening sight or optic nerve compression. The outcome of "stable" is defined if the ophthalmic outcome does not fit the definition of "improvement" or "deterioration".

SECONDARY OUTCOMES:
The change of quality of life (GO-QoL) | at 24 weeks and 48 weeks
  The outcome is grading as improvement, stable and deterioration. Improvement is defined if there are more than 6 points increase in any of the category in GO-QoL. Deterioration is defined if there are more than 6 points decrease in any of the category in GO-QoL. Stable is defined if none of above criteria is achieved.
The change of muscle volume (cm^3) on computed tomography | at 24 weeks and 48 weeks
  Change of muscle volume on noncontrast orbital CT
The change of fat volume (cm^3) on computed tomography | at 24 weeks and 48 weeks
  Change of fat volume on noncontrast orbital CT
The change of orbital volume (cm^3) on computed tomography | at 24 weeks and 48 weeks
  Change of orbital volume on noncontrast orbital CT
The change of muscle density on computed tomography | at 24 weeks and 48 weeks
  The density of muscle is measured and recorded in Hounsfield units.
The change of fat density on computed tomography | at 24 weeks and 48 weeks
  The density of fat is measured and recorded in Hounsfield units.
The change of diplopia score | at 24 weeks and 48 weeks
  The Gorman diplopia score includes four categories: no diplopia(absent), diplopia when the patient is tired or awakening (intermittent), diplopia at extremes of gaze (inconstant), and continuous diplopia in the primary or reading position (constant).
The change of clinical activity score (CAS) | at 24 weeks and 48 weeks
  Clinical activity score (CAS) is a 7-point scale using to evaluate the activity of GO in each eye. It includes 7 items to be scored respectively in each eye with minimum 0 point and maximum 7 points. More points indicate that GO in the eye is more active. The 7 items are listed as below:
  1. Spontaneous orbital pain
  2. Gaze evoked orbital pain
  3. Eyelid swelling that is considered to be due to active GO
  4. Eyelid erythema
  5. Conjunctival redness that is considered to be due to active GO
  6. Chemosis
  7. Inflammation of caruncle OR plica
The change of visual acuity | at 24 weeks and 48 weeks
  Evaluation of visual acuity will be done by the same ophthalmologist
The change of antithyroid peroxidase antibody (anti-TPO) (IU/mL) | at 24 weeks and 48 weeks
  Change of thyroid autoantibodies
The change of thyroglobulin antibody (TA) (IU/mL) | at 24 weeks and 48 weeks
  Change of thyroid autoantibodies
The change of thyrotropin-binding inhibiting immunoglobulin (TBII) (%). | at 24 weeks and 48 weeks
  Change of thyroid autoantibodies

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Hsin-Chu branch, Hsinchu
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) sharing is available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available after completed study enrollment.
Access Criteria: Individual participant data (IPD) sharing is available upon request.

REFERENCES:
- [Derived] Lin CH, Wei YH, Lu JY, Li HY, Lee CW, Yang CY, Chang CH, Wu WC, Wang CY, Shih SR. A randomized controlled trial on the effect of hydroxychloroquine in mild Graves' orbitopathy (GO-HCQ): study protocol. Trials. 2025 Aug 4;26(1):272. doi: 10.1186/s13063-025-09002-6. PMID 40760017